CLINICAL TRIAL: NCT01285167
Title: Daxas for COPD Therapy (DACOTA)
Brief Title: Quality of Life in Daxas-treated Patients Older Than 18 Years With Severe Chronic Obstructive Pulmonary Disease (COPD) (DACOTA)
Acronym: DACOTA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-401-DE; U1111-1136-8784 (Other: WHO)
Record Dates: First submitted 2011-01-21; First posted 2011-01-27 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Quality of life; lung function; spirometry; roflumilast; Daxas; severe COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DACOTA
  Interventions: Drug: Daxas

INTERVENTIONS:
Drug: Daxas — 500 microgram, oral, once daily as add-on therapy to existing therapy

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a progressive and largely irreversible lung disease characterized by chronic bronchitis and/or emphysema, resulting in breathlessness, cough and sputum. As COPD progresses, patients experience increasing deterioration of their health-related quality of life, with greater impairment in their ability to work and declining participation in social and physical activities.

The aim of this non-interventional study is to evaluate data on quality of life in COPD patients in Germany in a real life medical setting under therapy with the phosphodiesterase-inhibitor (PDE-4) roflumilast (Daxas). Evaluation is based on two COPD specific questionnaires to assess the patient's health status over six months. During the study, lung function measurements such as spirometry will be conducted according to common medical standard. Daxas (tablet) will be administered once daily. The study will provide further data on the safety and tolerability of Daxas.

ELIGIBILITY:
Main Inclusion Criteria:

* severe COPD

Main Exclusion Criteria:

* Child pugh (classified B and C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with severe COPD.
Sampling Method: Non-Probability Sample
Enrollment: 3645 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pre-/post comparison of the COPD status based on patients health status | after 6 months
  Evaluation of treatment success by a COPD-specific patient questionnaire

SECONDARY OUTCOMES:
Effectiveness during treatment | after 6 months
  Evaluation of treatment success by a health status patient questionnaire
Pre-/post comparison of spirometry data | after 6 months
Evaluation of tolerability | after 6 months
  assessment of adverse drug reactions
Evaluation of symptom reduction of sputum and cough | after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (447):
- Germany (447):
  - Nycomed Deutschland GmbH, Ahlen
  - Nycomed Deutschland GmbH, Allendorf
  - Nycomed Deutschland GmbH, Allersberg
  - Nycomed Deutschland GmbH, Alpenrod
  - Nycomed Deutschland GmbH, Altena
  - Nycomed Deutschland GmbH, Altenburg
  - Nycomed Deutschland GmbH, Alzenau in Unterfranken
  - Nycomed Deutschland GmbH, Alzey
  - Nycomed Deutschland GmbH, Amberg
  - Nycomed Deutschland GmbH, Anklam
  - Nycomed Deutschland GmbH, Annaberg-Buchholz
  - Nycomed Deutschland GmbH, Arnsberg
  - Nycomed Deutschland GmbH, Aschaffenburg
  - Nycomed Deutschland GmbH, Attendorn
  - Nycomed Deutschland GmbH, Attenkirchen
  - Nycomed Deutschland GmbH, Auerbach
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Backnang
  - Nycomed Deutschland GmbH, Bad Doberan
  - Nycomed Deutschland GmbH, Bad Endorf
  - Nycomed Deutschland GmbH, Bad Essen
  - Nycomed Deutschland GmbH, Bad Freienwalde
  - Nycomed Deutschland GmbH, Bad Füssing
  - Nycomed Deutschland GmbH, Bad Honnef
  - Nycomed Deutschland GmbH, Bad Langensalza
  - Nycomed Deutschland GmbH, Bad Lippspringe
  - Nycomed Deutschland GmbH, Bad Reichenhall
  - Nycomed Deutschland GmbH, Bad Salzuflen
  - Nycomed Deutschland GmbH, Bad Salzungen
  - Nycomed Deutschland GmbH, Bad Soden
  - Nycomed Deutschland GmbH, Bad Soden-Salmünster
  - Nycomed Deutschland GmbH, Bad Tennstedt
  - Nycomed Deutschland GmbH, Bad Wörishofen
  - Nycomed Deutschland GmbH, Badel
  - Nycomed Deutschland GmbH, Baden-Baden
  - Nycomed Deutschland GmbH, Bamberg
  - Nycomed Deutschland GmbH, Bargteheide
  - Nycomed Deutschland GmbH, Baunatal
  - Nycomed Deutschland GmbH, Bausendorf
  - Nycomed Deutschland GmbH, Bautzen
  - Nycomed Deutschland GmbH, Beelitz
  - Nycomed Deutschland GmbH, Bensheim
  - Nycomed Deutschland GmbH, Bergisch Gladbach
  - Nycomed Deutschland GmbH, Bergkamen
  - Nycomed Deutschland GmbH, Bergneustadt
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bernau
  - Nycomed Deutschland GmbH, Biedenkopf
  - Nycomed Deutschland GmbH, Bielefeld
  - Nycomed Deutschland GmbH, Bietigheim-Bissingen
  - Nycomed Deutschland GmbH, Bitterfeld-Wolfen
  - Nycomed Deutschland GmbH, Blankenhain
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bondorf
  - Nycomed Deutschland GmbH, Bonn
  - Nycomed Deutschland GmbH, Bonndorf
  - Nycomed Deutschland GmbH, Bottrop
  - Nycomed Deutschland GmbH, Bovenden
  - Nycomed Deutschland GmbH, Braunfels
  - Nycomed Deutschland GmbH, Braunsbedra
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Bredstedt
  - Nycomed Deutschland GmbH, Breitengüßbach
  - Nycomed Deutschland GmbH, Bremerhaven
  - Nycomed Deutschland GmbH, Brilon
  - Nycomed Deutschland GmbH, Bruchsal
  - Nycomed Deutschland GmbH, Brunsbüttel
  - Nycomed Deutschland GmbH, Buckow
  - Nycomed Deutschland GmbH, Burgau
  - Nycomed Deutschland GmbH, Burgstädt
  - Nycomed Deutschland GmbH, Burgwedel
  - Nycomed Deutschland GmbH, Büchen
  - Nycomed Deutschland GmbH, Büddenstedt
  - Nycomed Deutschland GmbH, Bünde
  - Nycomed Deutschland GmbH, Callenberg
  - Nycomed Deutschland GmbH, Camburg
  - Nycomed Deutschland GmbH, Celle
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Coburg
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Crimmitschau
  - Nycomed Deutschland GmbH, Darmstadt
  - Nycomed Deutschland GmbH, Deggendorf
  - Nycomed Deutschland GmbH, Deggingen
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Dillingen
  - Nycomed Deutschland GmbH, Dinslaken
  - Nycomed Deutschland GmbH, Dommitzsch
  - Nycomed Deutschland GmbH, Dornstetten
  - Nycomed Deutschland GmbH, Dorsten
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Dörentrup
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Duisburg
  - Nycomed Deutschland GmbH, Düren
  - Nycomed Deutschland GmbH, Düsseldorf
  - Nycomed Deutschland GmbH, Eberswalde
  - Nycomed Deutschland GmbH, Eggenfelden
  - Nycomed Deutschland GmbH, Ehra-Lessien
  - Nycomed Deutschland GmbH, Ehrenkirchen
  - Nycomed Deutschland GmbH, Einbeck
  - Nycomed Deutschland GmbH, Eisenach
  - Nycomed Deutschland GmbH, Ellerstadt
  - Nycomed Deutschland GmbH, Ellrich
  - Nycomed Deutschland GmbH, Ellwangen (Jagst)
  - Nycomed Deutschland GmbH, Emsdetten
  - Nycomed Deutschland GmbH, Emskirchen
  - Nycomed Deutschland GmbH, Ennepetal
  - Nycomed Deutschland GmbH, Erfde
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Erlangen
  - Nycomed Deutschland GmbH, Eschau
  - Nycomed Deutschland GmbH, Eschwege
  - Nycomed Deutschland GmbH, Eschweiler
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Essenheim
  - Nycomed Deutschland GmbH, Esslingen am Neckar
  - Nycomed Deutschland GmbH, Ettlingen
  - Nycomed Deutschland GmbH, Eutin
  - Nycomed Deutschland GmbH, Falkensee
  - Nycomed Deutschland GmbH, Feldberger Seenlandschaft
  - Nycomed Deutschland GmbH, Flensburg
  - Nycomed Deutschland GmbH, Flöha
  - Nycomed Deutschland GmbH, Frankenthal
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Frankfurt am Main
  - Nycomed Deutschland GmbH, Freising
  - Nycomed Deutschland GmbH, Friedrichshafen
  - Nycomed Deutschland GmbH, Fulda
  - Nycomed Deutschland GmbH, Fürstenfeldbruck
  - Nycomed Deutschland GmbH, Fürstenwalde
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Ganderkesee
  - Nycomed Deutschland GmbH, Gardelegen
  - Nycomed Deutschland GmbH, Garmisch-Partenkirchen
  - Nycomed Deutschland GmbH, Gauting
  - Nycomed Deutschland GmbH, Gelsenkirchen
  - Nycomed Deutschland GmbH, Gemünden
  - Nycomed Deutschland GmbH, Germering
  - Nycomed Deutschland GmbH, Gifhorn
  - Nycomed Deutschland GmbH, Gladbeck
  - Nycomed Deutschland GmbH, Glauchau
  - Nycomed Deutschland GmbH, Goch
  - Nycomed Deutschland GmbH, Gotha
  - Nycomed Deutschland GmbH, Gräfenhainichen
  - Nycomed Deutschland GmbH, Grebenstein
  - Nycomed Deutschland GmbH, Grefrath
  - Nycomed Deutschland GmbH, Greiz
  - Nycomed Deutschland GmbH, Grimmen
  - Nycomed Deutschland GmbH, Groß Kreutz
  - Nycomed Deutschland GmbH, Großaitingen
  - Nycomed Deutschland GmbH, Großefehn
  - Nycomed Deutschland GmbH, Großkorbetha
  - Nycomed Deutschland GmbH, Großschirma
  - Nycomed Deutschland GmbH, Grömitz
  - Nycomed Deutschland GmbH, Gütersloh
  - Nycomed Deutschland GmbH, Hagen
  - Nycomed Deutschland GmbH, Haibach
  - Nycomed Deutschland GmbH, Halbe
  - Nycomed Deutschland GmbH, Halberstadt
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Halstenbek
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hammelburg
  - Nycomed Deutschland GmbH, Hannoversch Münden
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Haren
  - Nycomed Deutschland GmbH, Hartha
  - Nycomed Deutschland GmbH, Haselünne
  - Nycomed Deutschland GmbH, Haßloch
  - Nycomed Deutschland GmbH, Heidelberg
  - Nycomed Deutschland GmbH, Heilbronn
  - Nycomed Deutschland GmbH, Heiligenhafen
  - Nycomed Deutschland GmbH, Heiligenhaus
  - Nycomed Deutschland GmbH, Heimbuchenthal
  - Nycomed Deutschland GmbH, Hemmingen
  - Nycomed Deutschland GmbH, Herbsleben
  - Nycomed Deutschland GmbH, Herne
  - Nycomed Deutschland GmbH, Herzlake
  - Nycomed Deutschland GmbH, Hettstedt
  - Nycomed Deutschland GmbH, Hille
  - Nycomed Deutschland GmbH, Hohenmölsen
  - Nycomed Deutschland GmbH, Homberg (Ohm)
  - Nycomed Deutschland GmbH, Homburg
  - Nycomed Deutschland GmbH, Horb
  - Nycomed Deutschland GmbH, Hoyerswerda
  - Nycomed Deutschland GmbH, Höchstadt an der Aisch
  - Nycomed Deutschland GmbH, Ibbenbueren
  - Nycomed Deutschland GmbH, Idstein
  - Nycomed Deutschland GmbH, Illerrieden
  - Nycomed Deutschland GmbH, Iserlohn
  - Nycomed Deutschland GmbH, Issum
  - Nycomed Deutschland GmbH, Itzehoe
  - Nycomed Deutschland GmbH, Jessen
  - Nycomed Deutschland GmbH, Jettingen
  - Nycomed Deutschland GmbH, Johannesberg
  - Nycomed Deutschland GmbH, Jübek
  - Nycomed Deutschland GmbH, Kaiserslautern
  - Nycomed Deutschland GmbH, Kalawa
  - Nycomed Deutschland GmbH, Kamen
  - Nycomed Deutschland GmbH, Kamenz
  - Nycomed Deutschland GmbH, Kandern
  - Nycomed Deutschland GmbH, Karlsruhe
  - Nycomed Deutschland GmbH, Kempten
  - Nycomed Deutschland GmbH, Kevelaer
  - Nycomed Deutschland GmbH, Kirchenlamitz
  - Nycomed Deutschland GmbH, Kirchheim
  - Nycomed Deutschland GmbH, Kleinostheim
  - Nycomed Deutschland GmbH, Klingenberg
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Konstanz
  - Nycomed Deutschland GmbH, Kornwestheim
  - Nycomed Deutschland GmbH, Königs Wusterhausen
  - Nycomed Deutschland GmbH, Köthen
  - Nycomed Deutschland GmbH, Krefeld
  - Nycomed Deutschland GmbH, Krumbach
  - Nycomed Deutschland GmbH, Krummhörn
  - Nycomed Deutschland GmbH, Kyritz
  - Nycomed Deutschland GmbH, Laage
  - Nycomed Deutschland GmbH, Lahr
  - Nycomed Deutschland GmbH, Lambrecht
  - Nycomed Deutschland GmbH, Landshut
  - Nycomed Deutschland GmbH, Langenfeld
  - Nycomed Deutschland GmbH, Langenhagen
  - Nycomed Deutschland GmbH, Langwedel
  - Nycomed Deutschland GmbH, Lathen
  - Nycomed Deutschland GmbH, Laubach
  - Nycomed Deutschland GmbH, Lehre
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Lensahn
  - Nycomed Deutschland GmbH, Leonberg
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Lichtenfels
  - Nycomed Deutschland GmbH, Limbach-Oberfrohna
  - Nycomed Deutschland GmbH, Limburg
  - Nycomed Deutschland GmbH, Lindenfels
  - Nycomed Deutschland GmbH, Lippetal
  - Nycomed Deutschland GmbH, Lippstadt
  - Nycomed Deutschland GmbH, Löbau
  - Nycomed Deutschland GmbH, Löhne
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Ludwigslust
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Lühmannsdorf
  - Nycomed Deutschland GmbH, Lüneburg
  - Nycomed Deutschland GmbH, Lützen
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Marienhafe
  - Nycomed Deutschland GmbH, Marienheide
  - Nycomed Deutschland GmbH, Marl
  - Nycomed Deutschland GmbH, Meckenbeuren
  - Nycomed Deutschland GmbH, Meckenheim
  - Nycomed Deutschland GmbH, Meerbusch
  - Nycomed Deutschland GmbH, Meisenheim
  - Nycomed Deutschland GmbH, Menden
  - Nycomed Deutschland GmbH, Mendig
  - Nycomed Deutschland GmbH, Merchweiler
  - Nycomed Deutschland GmbH, Merseburg
  - Nycomed Deutschland GmbH, Mertendorf
  - Nycomed Deutschland GmbH, Meuselwitz
  - Nycomed Deutschland GmbH, Miesbach
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, Moers
  - Nycomed Deutschland GmbH, Monheim
  - Nycomed Deutschland GmbH, Moormerland
  - Nycomed Deutschland GmbH, Mönchengladbach
  - Nycomed Deutschland GmbH, Mülheim
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münster
  - Nycomed Deutschland GmbH, Münzenberg
  - Nycomed Deutschland GmbH, Nauen
  - Nycomed Deutschland GmbH, Neckartailfingen
  - Nycomed Deutschland GmbH, Nettersheim
  - Nycomed Deutschland GmbH, Neuhausen
  - Nycomed Deutschland GmbH, Neumarkt
  - Nycomed Deutschland GmbH, Neunkirchen
  - Nycomed Deutschland GmbH, Neuss
  - Nycomed Deutschland GmbH, Neustadt
  - Nycomed Deutschland GmbH, Neuwied
  - Nycomed Deutschland GmbH, Nienburg
  - Nycomed Deutschland GmbH, Nordstemmen
  - Nycomed Deutschland GmbH, Nossen
  - Nycomed Deutschland GmbH, Nuremberg
  - Nycomed Deutschland GmbH, Obernzenn
  - Nycomed Deutschland GmbH, Oberursel
  - Nycomed Deutschland GmbH, Oer-Erkenschwick
  - Nycomed Deutschland GmbH, Offenbach
  - Nycomed Deutschland GmbH, Offenburg
  - Nycomed Deutschland GmbH, Oranienburg
  - Nycomed Deutschland GmbH, Ornbau
  - Nycomed Deutschland GmbH, Oschatz
  - Nycomed Deutschland GmbH, Oschersleben
  - Nycomed Deutschland GmbH, Osnabrück
  - Nycomed Deutschland GmbH, Osterode
  - Nycomed Deutschland GmbH, Ostrhauderfehn
  - Nycomed Deutschland GmbH, Paderborn
  - Nycomed Deutschland GmbH, Papenburg
  - Nycomed Deutschland GmbH, Parchim
  - Nycomed Deutschland GmbH, Pforzheim
  - Nycomed Deutschland GmbH, Pinneberg
  - Nycomed Deutschland GmbH, Pirmasens
  - Nycomed Deutschland GmbH, Plauen
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Pottenstein
  - Nycomed Deutschland GmbH, Radebeul
  - Nycomed Deutschland GmbH, Radevormwald
  - Nycomed Deutschland GmbH, Rain
  - Nycomed Deutschland GmbH, Rathenow
  - Nycomed Deutschland GmbH, Ratingen
  - Nycomed Deutschland GmbH, Raubach
  - Nycomed Deutschland GmbH, Recke
  - Nycomed Deutschland GmbH, Recklinghausen
  - Nycomed Deutschland GmbH, Regensburg
  - Nycomed Deutschland GmbH, Reichenbach
  - Nycomed Deutschland GmbH, Reichenschwand
  - Nycomed Deutschland GmbH, Remscheid
  - Nycomed Deutschland GmbH, Remse
  - Nycomed Deutschland GmbH, Rendsburg
  - Nycomed Deutschland GmbH, Rheine
  - Nycomed Deutschland GmbH, Rhinow
  - Nycomed Deutschland GmbH, Riesa
  - Nycomed Deutschland GmbH, Rieschweiler-Mühlbach
  - Nycomed Deutschland GmbH, Rodenbach
  - Nycomed Deutschland GmbH, Roetgen
  - Nycomed Deutschland GmbH, Roggenburg
  - Nycomed Deutschland GmbH, Rosenfeld
  - Nycomed Deutschland GmbH, Rosengarten
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Roth
  - Nycomed Deutschland GmbH, Rottach-Egern
  - Nycomed Deutschland GmbH, Rödermark
  - Nycomed Deutschland GmbH, Rudolstadt
  - Nycomed Deutschland GmbH, Rüsselsheim am Main
  - Nycomed Deutschland GmbH, Saal
  - Nycomed Deutschland GmbH, Saalfeld
  - Nycomed Deutschland GmbH, Saarbrücken
  - Nycomed Deutschland GmbH, Saarlouis
  - Nycomed Deutschland GmbH, Sachsenheim
  - Nycomed Deutschland GmbH, Saint Blasien
  - Nycomed Deutschland GmbH, Salzmünde
  - Nycomed Deutschland GmbH, Schieder-Schwalenberg
  - Nycomed Deutschland GmbH, Schloß Holte-Stukenbrock
  - Nycomed Deutschland GmbH, Schlüchtern
  - Nycomed Deutschland GmbH, Schmölln
  - Nycomed Deutschland GmbH, Schönberg
  - Nycomed Deutschland GmbH, Schönebeck
  - Nycomed Deutschland GmbH, Schrobenhausen
  - Nycomed Deutschland GmbH, Schwalbach
  - Nycomed Deutschland GmbH, Schwalmstadt
  - Nycomed Deutschland GmbH, Schwanewede
  - Nycomed Deutschland GmbH, Schwäbisch Gmünd
  - Nycomed Deutschland GmbH, Schwedt
  - Nycomed Deutschland GmbH, Schweinfurt
  - Nycomed Deutschland GmbH, Schwerin
  - Nycomed Deutschland GmbH, Schwetzingen
  - Nycomed Deutschland GmbH, Sebnitz
  - Nycomed Deutschland GmbH, Seelow
  - Nycomed Deutschland GmbH, Seevetal
  - Nycomed Deutschland GmbH, Seewald
  - Nycomed Deutschland GmbH, Sendenhorst
  - Nycomed Deutschland GmbH, Sickte
  - Nycomed Deutschland GmbH, Siegen
  - Nycomed Deutschland GmbH, Simmern
  - Nycomed Deutschland GmbH, Simmertal
  - Nycomed Deutschland GmbH, Sinntal
  - Nycomed Deutschland GmbH, Sinsheim
  - Nycomed Deutschland GmbH, Solingen
  - Nycomed Deutschland GmbH, Soltau
  - Nycomed Deutschland GmbH, Sonneberg
  - Nycomed Deutschland GmbH, Sömmerda
  - Nycomed Deutschland GmbH, Speyer
  - Nycomed Deutschland GmbH, Sprockhövel
  - Nycomed Deutschland GmbH, Stadtallendorf
  - Nycomed Deutschland GmbH, Stadthagen
  - Nycomed Deutschland GmbH, Staig
  - Nycomed Deutschland GmbH, Steimel
  - Nycomed Deutschland GmbH, Steinbach
  - Nycomed Deutschland GmbH, Steinfeld
  - Nycomed Deutschland GmbH, Steinhagen
  - Nycomed Deutschland GmbH, Stockach
  - Nycomed Deutschland GmbH, Straelen
  - Nycomed Deutschland GmbH, Stralsund
  - Nycomed Deutschland GmbH, Straupitz
  - Nycomed Deutschland GmbH, Strausberg
  - Nycomed Deutschland GmbH, Stuhr
  - Nycomed Deutschland GmbH, Stuttgart
  - Nycomed Deutschland GmbH, Sundern
  - Nycomed Deutschland GmbH, Sülz
  - Nycomed Deutschland GmbH, Süßen
  - Nycomed Deutschland GmbH, Tangermünde
  - Nycomed Deutschland GmbH, Teltow
  - Nycomed Deutschland GmbH, Teterow
  - Nycomed Deutschland GmbH, Teuchern
  - Nycomed Deutschland GmbH, Teutschenthal
  - Nycomed Deutschland GmbH, Thurnau
  - Nycomed Deutschland GmbH, Tirschenreuth
  - Nycomed Deutschland GmbH, Tuttlingen
  - Nycomed Deutschland GmbH, Uchte
  - Nycomed Deutschland GmbH, Ueckermünde
  - Nycomed Deutschland GmbH, Ulm
  - Nycomed Deutschland GmbH, Unna
  - Nycomed Deutschland GmbH, Urbach
  - Nycomed Deutschland GmbH, Uttenreuth
  - Nycomed Deutschland GmbH, Überlingen
  - Nycomed Deutschland GmbH, Vaihingen
  - Nycomed Deutschland GmbH, Viersen
  - Nycomed Deutschland GmbH, Villingen-Schwenningen
  - Nycomed Deutschland GmbH, Vilshofen
  - Nycomed Deutschland GmbH, Voerde
  - Nycomed Deutschland GmbH, Waiblingen
  - Nycomed Deutschland GmbH, Wandlitz
  - Nycomed Deutschland GmbH, Waren
  - Nycomed Deutschland GmbH, Weidenberg
  - Nycomed Deutschland GmbH, Weilheim
  - Nycomed Deutschland GmbH, Weißenfels
  - Nycomed Deutschland GmbH, Weißwasser
  - Nycomed Deutschland GmbH, Werder
  - Nycomed Deutschland GmbH, Wetter
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wiesloch
  - Nycomed Deutschland GmbH, Wilhermsdorf
  - Nycomed Deutschland GmbH, Wilster
  - Nycomed Deutschland GmbH, Winhöring
  - Nycomed Deutschland GmbH, Wissen
  - Nycomed Deutschland GmbH, Witten
  - Nycomed Deutschland GmbH, Wittenberg
  - Nycomed Deutschland GmbH, Wittislingen
  - Nycomed Deutschland GmbH, Wittstock
  - Nycomed Deutschland GmbH, Wolfsburg
  - Nycomed Deutschland GmbH, Wolfschlugen
  - Nycomed Deutschland GmbH, Wolgast
  - Nycomed Deutschland GmbH, Wöllstein
  - Nycomed Deutschland GmbH, Wörth
  - Nycomed Deutschland GmbH, Wulfen
  - Nycomed Deutschland GmbH, Würzburg
  - Nycomed Deutschland GmbH, Wyhl
  - Nycomed Deutschland GmbH, Xanten
  - Nycomed Deutschland GmbH, Zeitz
  - Nycomed Deutschland GmbH, Zellingen
  - Nycomed Deutschland GmbH, Zerbst
  - Nycomed Deutschland GmbH, Zossen
  - Nycomed Deutschland GmbH, Zühlsdorf
  - Nycomed Deutschland GmbH, Zwickau